CLINICAL TRIAL: NCT03871062
Title: A Prospective, Randomised, Single-masked Comparison of Topical Anesthesia and Topical Combined Subconjunctival (Two-step) Anesthesia in Intravitreal Injection
Brief Title: Study of Two-step Anesthesia in Intravitreal Injection
Acronym: TAIVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SHIRB20190228
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, Local
Keywords: intravitreal injection; pain; anesthesia
MeSH Terms: conditions — Pain | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical anesthesia group (Active Comparator): conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times
  Interventions: Procedure: topical anesthesia
- two step anesthesia group (Experimental): conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times + 2% lidocaine 0.2 ml subconjunctival injection
  Interventions: Procedure: Two step anesthesia

INTERVENTIONS:
Procedure: Two step anesthesia — conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times + 2% lidocaine 0.2 ml subconjunctival injection
  Arms: two step anesthesia group
Procedure: topical anesthesia — conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times
  Arms: topical anesthesia group

SUMMARY:
A prospective, randomised, single-masked comparison of local anaesthetic approaches including topical anesthesia combined sub-conjunctival anesthesia (two-step anesthesia) for intravitreal injection #TAIVI# vs topical anesthesia

DETAILED DESCRIPTION:
Purpose: Patient pain for intravitreal injection is evaluated between topical anesthesia combined sub-conjunctival anesthesia (two-step anesthesia) and topical anesthesia.

Methods: This prospective, randomized, single-blinded clinical trail is conducted at Shanghai Aier Eye Hospital. Selected group of 60 patients will be randomized divided into 2 groups and underwent intravitreal injection of antiangiogenic agents and steroids. Group1 uses two-step anesthesia , whereas Group 2 uses topical anesthesia. A 5-point Visual Analogue Pain Scale is used to assess patients' pain score and surgeon's ease while operating. Any complications therefore will be made note of.

ELIGIBILITY:
Inclusion Criteria:

Neovascular age-related macular degeneration (wAMD); Pathologic myopia with choroidal neovascularisation (PM-CNV); Diabetic macular edema (DME); Retinal vein occlusion with macular edema (RVO-ME); Other diseases: uveitis with macular edema or choroidal neovascularisation.

Exclusion Criteria:

Communication problems; Allergy to amide-type local anaesthetic agents; History of vitreoretinal surgery or orbital surgery; Orbital deformity; With episcleral adjunct surgery; Trauma; Keratitis; Conjunctivitis.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-08 (Estimated); Primary Completion 2019-09-11 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores | During surgery
  5-point Visual Analogue Pain Scale (VAPS): Grade 1: No pain or discomfort; Grade 2: mild pain or discomfort; Grade 3: moderate pain or discomfort; Grade 4: severe pain or discomfort

SECONDARY OUTCOMES:
Surgeon's ease | During surgery
  Grade 1: No discomfort; Grade 2: mild discomfort; Grade 3: moderate discomfort; Grade 4: severe discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Study Director — Shanghai Aier Eye Hosptial
Locations (1):
- Shanghai Aier Eye Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shiroma HF, Takaschima AKK, Farah ME, Hofling-Lima AL, de Luca Canto G, Benedetti RH, Rodrigues EB. Patient pain during intravitreal injections under topical anesthesia: a systematic review. Int J Retina Vitreous. 2017 Jul 3;3:23. doi: 10.1186/s40942-017-0076-9. eCollection 2017. PMID 28680703
- [Result] Blaha GR, Tilton EP, Barouch FC, Marx JL. Randomized trial of anesthetic methods for intravitreal injections. Retina. 2011 Mar;31(3):535-9. doi: 10.1097/IAE.0b013e3181eac724. PMID 21102369
- [Result] Shin SH, Park SP, Kim YK. Factors Associated with Pain Following Intravitreal Injections. Korean J Ophthalmol. 2018 Jun;32(3):196-203. doi: 10.3341/kjo.2017.0081. Epub 2018 May 15. PMID 29770638
- [Result] Nguyen NCI, Fabro F, Ambresin A, Ezziat S, Bergin C, Mazzocato C, Mantel I. Factors associated with pain during intravitreal injection of anti-vascular endothelial growth factor. Eye (Lond). 2018 Sep;32(9):1544-1546. doi: 10.1038/s41433-018-0126-z. Epub 2018 May 17. No abstract available. PMID 29769650
- [Result] Sanabria MR, Montero JA, Losada MV, Fernandez-Munoz M, Galindo A, Fernandez I, Coco RM, Sampedro A. Ocular pain after intravitreal injection. Curr Eye Res. 2013 Feb;38(2):278-82. doi: 10.3109/02713683.2012.758290. Epub 2013 Jan 18. PMID 23330822